CLINICAL TRIAL: NCT00625378
Title: Sorafenib Long Term Extension Program
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12311; 2007-002604-17 (EudraCT Number)
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms
Keywords: Cancer; Sorafenib; Extension program
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Participants receive single-agent sorafenib at the same dose and schedule as in their original clinical trials.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — At the same dose and schedule as in the participants' original clinical trials

SUMMARY:
The primary purpose of program was to enable patients, currently receiving sorafenib (Nexavar) in a Bayer/Onyx sponsored clinical trial, to continue sorafenib treatment after their respective study had met its primary endpoint and/or had reached the end as defined in the original protocol. Patients were able to continue treatment until (i) the treating physician felt the patient was no longer benefiting from the treatment or (ii) the treatment becomes commercially available and reimbursed for the respective indication as applicable in the country in which the patient lived and the patient could obtain suitable amounts of drug for treatment through standard mechanisms of commercial availability (ie, there should be no interruption in the patient's treatment schedule when switching to commercially available product) or (iii) the patient could join a Post-Trial-Access Program, another study or can receive sorafenib through any other mechanism (e.g. local access program) in accordance with local legal and compliance rules, with no cost to the patient with respect to sorafenib.

An additional objective was the assessment of the safety of Nexavar or Nexavar combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who are participating in a previous Bayer/Onyx sponsored study that has reached its endpoint (statistical and regulatory or study end), and who are, in the opinion of the Investigator, expected to continue to have an overall positive benefit/risk from continuing treatment.
* Patients who have signed informed consent for this long term extension program.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 days period after last study drug dosing. The investigator should advise the patient how to achieve an adequate contraception.
* Women of childbearing potential who have a negative pregnancy test within 7 days of the first dose of sorafenib in this long term extension program.
* Patient is receiving sorafenib (Nexavar) as a monotherapy in their originating protocol. Patients who were being treated with sorafenib (Nexavar) in combination with other chemotherapies in the original study, but continued on single agent sorafenib (Nexavar) after discontinuation of the combination agent will be eligible.
* Patient who are receiving concurrent combination with sorafenib (Nexavar) and TACE (transarterial chemoembolization) in their originating study will be eligible.
* Patients who are receiving concurrent combination with sorafenib (Nexavar) and capecitabine in their originating Study 12444 (RESILIENCE) will be eligible.
* Patients who are receiving concurrent combination with sorafenib (Nexavar) and erlotinib in their originating study 12917 (SEARCH) were eligible.
* Patients who have completed the End of Treatment assessments in their originating study. Every effort should be made to conduct the End of Treatment visit such that the patient does not have any interruption of sorafenib dosing.

Exclusion Criteria:

* Any condition that is unstable or that could jeopardize the safety of the patient (please refer to the Investigator Brochure and product labeling safety sections).
* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class 2 or uncontrolled hypertension.
* Myocardial infarction (MI) within the last 3 months.
* Symptomatic metastatic brain or meningeal tumors .
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors ( Ta, Tis &T1) or any cancer curatively treated > 5 years prior to study entry.
* Patients with seizure disorder requiring medication (such as steroid anti-epileptics).
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Any condition which could jeopardise the safety of the patient and his/her compliance in the study.

Excluded therapies and medications, previous and concomitant:

* Concurrent anti-cancer chemotherapy, except transarterial chemoembolization (TACE) and capecitabine
* Concurrent immunotherapy (including monoclonal antibodies), during or within 30 days prior to start of study drug
* Concurrent hormonal therapy, except for bisphosphonates,during or within 30 days prior to start of study drug
* Concomitant Rifampicin and St John's Wort (Warfarin may be used only with very close monitoring)
* Radiotherapy during study or within 3 weeks of start of study drug. [Palliative radiotherapy will be allowed]
* Concomitant use of potent inhibitors of CYP3A4 including ketoconazole, itraconazole and ritonavir. Consumption of grapefruit juice should also be avoided.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-12-21 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- United States (4):
  - Los Angeles, California
  - New Haven, Connecticut
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
- Randwick, New South Wales, Australia
- Belgium (2):
  - Bruxelles - Brussel
  - Charleroi
- São Paulo, Brazil
- Bulgaria (2):
  - Plovdiv
  - Varna
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- China (5):
  - Guangzhou, Guangdong
  - Xi’an, Shanxi
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Floridablanca, Santander Department, Colombia
- Bordeaux, France
- Germany (6):
  - Gauting, Bavaria
  - Regensburg, Bavaria
  - Essen, North Rhine-Westphalia
  - Großhansdorf, Schleswig-Holstein
  - Berlin
  - Hamburg
- Hong Kong, Hong Kong
- Italy (8):
  - Bologna, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Milan, Lombardy
  - Pavia, Lombardy
  - Turin, Piedmont
  - Pisa, Tuscany
  - Siena, Tuscany
  - Perugia, Umbria
- Auckland, New Zealand
- Poland (5):
  - Gdansk
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
- South Korea (3):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Seoul
- Spain (5):
  - Oviedo, Principality of Asturias
  - Alicante
  - Barcelona
  - Madrid
  - Valencia
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Kiev, Ukraine
- United Kingdom (6):
  - Southampton, Hampshire
  - Maidstone, Kent
  - Cardiff, South Glamorgan
  - Sutton, Surrey
  - Glasgow
  - London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 19 countries between 21-Dec-2007 (first participant first visit) and 24-Sep-2021 (last participant last visit).
Pre-assignment Details: Overall, 206 participants were transferred from the feeder studies and have signed informed consent for STEP. Of these 206 participants, 2 participants were never treated and 204 participants received the study treatment.
Groups:
- Sorafenib Monotherapy: Participants received single-agent sorafenib at the same dose and schedule as in their original Clinical Trial.
- Sorafenib+Erlotinib: Participants received sorafenib and erlotinib combination at the same dose and schedule as in their original Clinical Trial.
Period: Overall Study
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Started | 205 | 1
Treated in STEP | 203 | 1
Completed | 0 | 0
Not Completed | 205 | 1
Not completed — Adverse Event | 22 | 0
Not completed — Withdrawal by Subject | 16 | 0
Not completed — Death | 38 | 0
Not completed — Disease progression, recurrence or relapse | 88 | 0
Not completed — Lost to Follow-up | 17 | 0
Not completed — Non-compliant with study medication | 3 | 0
Not completed — Investigator's judgement (no need to continue treatment) | 1 | 0
Not completed — Medical decision | 1 | 0
Not completed — Multiple toxicities | 1 | 0
Not completed — New cancer | 1 | 0
Not completed — PTA program | 2 | 0
Not completed — Recurrent rise in amylase and lipase | 1 | 0
Not completed — Sponsor decision | 1 | 0
Not completed — Sponsor's decision to stop the trial | 1 | 0
Not completed — Switch to commercial drug | 6 | 1
Not completed — Missing | 2 | 0
Not completed — End of treatment not available | 2 | 0
Not completed — Never treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF, included all participants who received at least one dose of study medication)
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib | Total
Number analyzed (Participants) | 203 | 1 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.6) | 20.0 (NA) — Value was not calculated due to the only 1 subject in the group | 63.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 0 | 63
  Male | 140 | 1 | 141
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 39 | 1 | 40
  Hispanic | 2 | 0 | 2
  Japanese/American | 1 | 0 | 1
  White | 161 | 0 | 161
ECOG performance status [Count of Participants; unit: Participants] — Eastern cooperative oncology group (ECOG) performance status: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours
  Participants
    ECOG 0 | 25 | 1 | 26
    ECOG 1 | 16 | 0 | 16
    ECOG 2 | 1 | 0 | 1
    Missing | 161 | 0 | 161

OUTCOME MEASURES:

1. Primary Outcome: Sorafenib Treatment Duration Within STEP
Description: Treatment duration was calculated in days as the date of the last dose of any study treatment minus date of the first dose of any study treatment plus one day.
Time Frame: From the date of the first sorafenib dose until the date of the last sorafenib dose, with a mean duration of 25 months and max duraton of 153.8 months
Population: Safety analysis set (SAF)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Months | 15.69 [6.41 to 33.19] | 40.13 [40.13 to 40.13]

2. Primary Outcome: Number of Participants With New Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The adverse event did not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death; was life-threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; was a congenital anomaly or birth defect; was an important medical event. A new treatment-emergent adverse event (TEAE) was any AE that had a start date on or after ICF date in STEP and up to 30 days after the last sorafenib dose. A drug-related new TEAE was any new TEAE that had a causal relationship with the study treatment as assessed by the investigator.
Time Frame: From signing the informed consent form (ICF) in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Any AE | 166 | 1
  Serious AE (SAE) | 113 | 1
  AE leading to dose modification | 64 | 0
  AE leading to study drug discontinuation | 56 | 0
  AE leading to death | 37 | 0
  Sorafenib-related AE | 117 | 1
  Sorafenib-related SAE | 25 | 1
  Sorafenib-related AE leading to dose modification | 42 | 0
  Sorafenib-related AE leading to study drug discontinuation | 21 | 0
  Sorafenib-related AE leading to death | 2 | 0

3. Primary Outcome: Number of Participants With New TEAEs of CTCAE Grades 3 or Higher by Worst CTCAE Grade
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The AE did not necessarily have to have a causal relationship with this treatment. A new treatment-emergent adverse event (TEAE) was any AE that had a start date on or after ICF date in STEP and up to 30 days after the last sorafenib dose. The intensity or severity of AEs were graded using the National Cancer Institute-Common Terminology Criteria, Version 3.0 (NCI-CTC v. 3.0). The Common Terminology Criteria for AE (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. It uses a range of grades from 1 to 5. Specific conditions and symptoms may have values or descriptive comment for each level, but the general guideline is: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe; Grade 4 - life-threatening; Grade 5 - death.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Grade 3 | 71 | 1
  Grade 4 | 17 | 1
  Grade 5 | 37 | 0

4. Primary Outcome: Number of Participants With Study Drug-related New TEAEs of CTCAE Grades 3 or Higher by Worst CTCAE Grade
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The AE did not necessarily have to have a causal relationship with this treatment. A new treatment-emergent AE (TEAE) was any AE that had a start date on or after ICF date in STEP and up to 30 days after the last sorafenib dose. A drug-related new TEAE was a new TEAE that had a causal relationship with the study treatment as assessed by the investigator. The intensity or severity of AEs were graded using the National Cancer Institute-Common Terminology Criteria (CTC v3). The Common Terminology Criteria for AE (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. It uses a range of grades from 1 to 5. The general guideline is: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe; Grade 4 - life-threatening; Grade 5 - death.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Grade 3 | 49 | 1
  Grade 4 | 6 | 0
  Grade 5 | 2 | 0

5. Primary Outcome: Number of Participants With All Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The AE did not necessarily have to have a causal relationship with this treatment. A drug-related AE was any AE that had a causal relationship with the study treatment as assessed by the investigator. All AEs in STEP were the combination of AEs ongoing from feeder studies and new TEAEs.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Any AE | 184 | 1
  Serious AE (SAE) | 114 | 1
  AE leading to dose modification | 72 | 0
  AE leading to study drug discontinuation | 56 | 0
  AE leading to death | 37 | 0
  Sorafenib-related AE | 159 | 1
  Sorafenib-related SAE | 26 | 1
  Sorafenib-related AE leading to dose modification | 53 | 0
  Sorafenib-related AE leading to study drug discontinuation | 21 | 0
  Sorafenib-related AE leading to death | 2 | 0

6. Primary Outcome: Number of Participants With All Adverse Events of CTCAE Grades 3 or Higher by Worst CTCAE Grade
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The AE did not necessarily have to have a causal relationship with this treatment. All AEs in STEP were the combination of AEs ongoing from feeder studies and new TEAEs. The intensity or severity of AEs were graded using the National Cancer Institute-Common Terminology Criteria, Version 3.0 (NCI-CTC v. 3.0). The Common Terminology Criteria for AE (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. It uses a range of grades from 1 to 5. Specific conditions and symptoms may have values or descriptive comment for each level, but the general guideline is: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe; Grade 4 - life-threatening; Grade 5 - death.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Grade 3 | 81 | 1
  Grade 4 | 17 | 1
  Grade 5 | 37 | 0

7. Primary Outcome: Number of Participants With Study Drug-related All Adverse Events of CTCAE Grades 3 or Higher by Worst CTCAE
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product. The AE did not necessarily have to have a causal relationship with this treatment. A drug-related AE was any AE that had a causal relationship with the study treatment as assessed by the investigator. All AEs in STEP was a combination of AEs ongoing from feeder studies and new TEAEs. The intensity or severity of AEs were graded using the National Cancer Institute-Common Terminology Criteria, Version 3.0 (NCI-CTC v. 3.0). The Common Terminology Criteria for AE (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. It uses a range of grades from 1 to 5. Specific conditions and symptoms may have values or descriptive comment for each level, but the general guideline is: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe; Grade 4 - life-threatening; Grade 5 - death.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Grade 3 | 65 | 1
  Grade 4 | 6 | 0
  Grade 5 | 2 | 0

8. Primary Outcome: Number of Deaths With Primary Cause of Death
Description: Primary cause of death included: any cause; progressive disease; toxicity due to study treatment (with at least one AE with outcome death); other (unspecified) or missing cause.
Time Frame: From signing the ICF in STEP until completion or discontinuation of the study, with a mean duration of 26 months
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Any cause | 62 | 0
  Progressive disease | 34 | 0
  Toxicity due to study treatment | 3 | 0
  Other | 21 | 0
  Missing | 4 | 0

9. Primary Outcome: Number of Participants With Abnormal Hematological and Biochemical Laboratory Values by Worst CTCAE Grade
Description: Hematology and blood chemistry values were summarized according to their worst CTCAE grade, where applicable. Hematology and blood chemistry values were graded based on the applicable laboratory threshold values outlined in NCI CTCAE version 3.0. Participants with a specific laboratory value that were "not graded" are not included in the table. CTCAE grade was set to "not graded" if the reference ranges or other information necessary to derive grades were unavailable or result had a special character (such as > or < ). The Common Terminology Criteria for Adverse Events (CTCAE) are a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. It uses a range of grades from 1 to 5. Specific conditions and symptoms may have values or descriptive comment for each level, but the general guideline is: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe; Grade 4 - life-threatening; Grade 5 - death.
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months
Population: Participants in safety analysis set (SAF) with evaluable data for each evaluated laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 203 | 1
Participants
  Neutrophils - Grade 1: number analyzed (Participants) | 165 | 0
  Neutrophils - Grade 1 | 19 |
  Neutrophils - Grade 2: number analyzed (Participants) | 165 | 0
  Neutrophils - Grade 2 | 7 |
  Neutrophils - Grade 3: number analyzed (Participants) | 165 | 0
  Neutrophils - Grade 3 | 0 |
  Neutrophils - Grade 4: number analyzed (Participants) | 165 | 0
  Neutrophils - Grade 4 | 2 |
  Hemoglobin - Grade 1: number analyzed (Participants) | 191 | 1
  Hemoglobin - Grade 1 | 67 | 1
  Hemoglobin - Grade 2: number analyzed (Participants) | 191 | 1
  Hemoglobin - Grade 2 | 40 | 0
  Hemoglobin - Grade 3: number analyzed (Participants) | 191 | 1
  Hemoglobin - Grade 3 | 13 | 0
  Hemoglobin - Grade 4: number analyzed (Participants) | 191 | 1
  Hemoglobin - Grade 4 | 8 | 0
  Lymphopenia - Grade 1: number analyzed (Participants) | 187 | 1
  Lymphopenia - Grade 1 | 37 | 0
  Lymphopenia - Grade 2: number analyzed (Participants) | 187 | 1
  Lymphopenia - Grade 2 | 37 | 0
  Lymphopenia - Grade 3: number analyzed (Participants) | 187 | 1
  Lymphopenia - Grade 3 | 20 | 0
  Lymphopenia - Grade 4: number analyzed (Participants) | 187 | 1
  Lymphopenia - Grade 4 | 4 | 1
  Platelets - Grade 1: number analyzed (Participants) | 189 | 1
  Platelets - Grade 1 | 48 | 0
  Platelets - Grade 2: number analyzed (Participants) | 189 | 1
  Platelets - Grade 2 | 7 | 0
  Platelets - Grade 3: number analyzed (Participants) | 189 | 1
  Platelets - Grade 3 | 7 | 0
  Platelets - Grade 4: number analyzed (Participants) | 189 | 1
  Platelets - Grade 4 | 17 | 1
  Leukocytes - Grade 1: number analyzed (Participants) | 192 | 1
  Leukocytes - Grade 1 | 40 | 1
  Leukocytes - Grade 2: number analyzed (Participants) | 192 | 1
  Leukocytes - Grade 2 | 12 | 0
  Leukocytes - Grade 3: number analyzed (Participants) | 192 | 1
  Leukocytes - Grade 3 | 2 | 0
  Leukocytes - Grade 4: number analyzed (Participants) | 192 | 1
  Leukocytes - Grade 4 | 1 | 0
  INR - Grade 1: number analyzed (Participants) | 82 | 0
  INR - Grade 1 | 17 |
  INR - Grade 2: number analyzed (Participants) | 82 | 0
  INR - Grade 2 | 1 |
  INR - Grade 3: number analyzed (Participants) | 82 | 0
  INR - Grade 3 | 11 |
  INR - Grade 4: number analyzed (Participants) | 82 | 0
  INR - Grade 4 | 0 |
  ALT - Grade 1: number analyzed (Participants) | 174 | 1
  ALT - Grade 1 | 66 | 1
  ALT - Grade 2: number analyzed (Participants) | 174 | 1
  ALT - Grade 2 | 13 | 0
  ALT - Grade 3: number analyzed (Participants) | 174 | 1
  ALT - Grade 3 | 7 | 0
  ALT - Grade 4: number analyzed (Participants) | 174 | 1
  ALT - Grade 4 | 0 | 0
  Amylase - Grade 1: number analyzed (Participants) | 178 | 1
  Amylase - Grade 1 | 39 | 1
  Amylase - Grade 2: number analyzed (Participants) | 178 | 1
  Amylase - Grade 2 | 12 | 0
  Amylase - Grade 3: number analyzed (Participants) | 178 | 1
  Amylase - Grade 3 | 8 | 0
  Amylase - Grade 4: number analyzed (Participants) | 178 | 1
  Amylase - Grade 4 | 0 | 0
  AST - Grade 1: number analyzed (Participants) | 183 | 1
  AST - Grade 1 | 88 | 1
  AST - Grade 2: number analyzed (Participants) | 183 | 1
  AST - Grade 2 | 19 | 0
  AST - Grade 3: number analyzed (Participants) | 183 | 1
  AST - Grade 3 | 6 | 0
  AST - Grade 4: number analyzed (Participants) | 183 | 1
  AST - Grade 4 | 0 | 0
  Lipase - Grade 1: number analyzed (Participants) | 165 | 1
  Lipase - Grade 1 | 32 | 0
  Lipase - Grade 2: number analyzed (Participants) | 165 | 1
  Lipase - Grade 2 | 11 | 1
  Lipase - Grade 3: number analyzed (Participants) | 165 | 1
  Lipase - Grade 3 | 28 | 0
  Lipase - Grade 4: number analyzed (Participants) | 165 | 1
  Lipase - Grade 4 | 7 | 0

10. Primary Outcome: Number of Participants With ECOG Performance Status by 6-months Time Intervals
Description: Eastern cooperative oncology group (ECOG) performance status: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5 = Dead
Time Frame: Up to 156 months
Population: Participants in safety analysis set (SAF) with evaluable data for the evaluation at each timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
Number analyzed (Participants) | 64 | 1
Participants
  Months 1-6: number analyzed (Participants) | 42 | 1
  Months 1-6: Missing | 2 | 0
  Months 1-6: ECOG 0 | 28 | 1
  Months 1-6: ECOG 1 | 11 | 0
  Months 1-6: ECOG 2 | 1 | 0
  Months 1-6: ECOG 3 | 0 | 0
  Months 1-6: ECOG 4 | 0 | 0
  Months 1-6: ECOG 5 | 0 | 0
  Months 7-12: number analyzed (Participants) | 38 | 1
  Months 7-12: Missing | 3 | 0
  Months 7-12: ECOG 0 | 29 | 1
  Months 7-12: ECOG 1 | 6 | 0
  Months 7-12: ECOG 2 | 0 | 0
  Months 7-12: ECOG 3 | 0 | 0
  Months 7-12: ECOG 4 | 0 | 0
  Months 7-12: ECOG 5 | 0 | 0
  Months 13-18: number analyzed (Participants) | 33 | 1
  Months 13-18: Missing | 2 | 0
  Months 13-18: ECOG 0 | 22 | 1
  Months 13-18: ECOG 1 | 7 | 0
  Months 13-18: ECOG 2 | 1 | 0
  Months 13-18: ECOG 3 | 1 | 0
  Months 13-18: ECOG 4 | 0 | 0
  Months 13-18: ECOG 5 | 0 | 0
  Months 19-24: number analyzed (Participants) | 28 | 1
  Months 19-24: Missing | 2 | 0
  Months 19-24: ECOG 0 | 15 | 1
  Months 19-24: ECOG 1 | 9 | 0
  Months 19-24: ECOG 2 | 1 | 0
  Months 19-24: ECOG 3 | 0 | 0
  Months 19-24: ECOG 4 | 0 | 0
  Months 19-24: ECOG 5 | 1 | 0
  Months 25-30: number analyzed (Participants) | 23 | 1
  Months 25-30: Missing | 2 | 0
  Months 25-30: ECOG 0 | 13 | 1
  Months 25-30: ECOG 1 | 7 | 0
  Months 25-30: ECOG 2 | 0 | 0
  Months 25-30: ECOG 3 | 0 | 0
  Months 25-30: ECOG 4 | 0 | 0
  Months 25-30: ECOG 5 | 1 | 0
  Months 31-36: number analyzed (Participants) | 19 | 1
  Months 31-36: Missing | 1 | 0
  Months 31-36: ECOG 0 | 9 | 1
  Months 31-36: ECOG 1 | 8 | 0
  Months 31-36: ECOG 2 | 0 | 0
  Months 31-36: ECOG 3 | 0 | 0
  Months 31-36: ECOG 4 | 0 | 0
  Months 31-36: ECOG 5 | 1 | 0
  Months 37-42: number analyzed (Participants) | 19 | 1
  Months 37-42: Missing | 0 | 0
  Months 37-42: ECOG 0 | 10 | 1
  Months 37-42: ECOG 1 | 8 | 0
  Months 37-42: ECOG 2 | 0 | 0
  Months 37-42: ECOG 3 | 0 | 0
  Months 37-42: ECOG 4 | 0 | 0
  Months 37-42: ECOG 5 | 1 | 0
  Months 43-48: number analyzed (Participants) | 16 | 0
  Months 43-48: Missing | 0 | 0
  Months 43-48: ECOG 0 | 9 | 0
  Months 43-48: ECOG 1 | 6 | 0
  Months 43-48: ECOG 2 | 0 | 0
  Months 43-48: ECOG 3 | 0 | 0
  Months 43-48: ECOG 4 | 0 | 0
  Months 43-48: ECOG 5 | 1 | 0
  Months 49-54: number analyzed (Participants) | 13 | 0
  Months 49-54: Missing | 0 | 0
  Months 49-54: ECOG 0 | 7 | 0
  Months 49-54: ECOG 1 | 6 | 0
  Months 49-54: ECOG 2 | 0 | 0
  Months 49-54: ECOG 3 | 0 | 0
  Months 49-54: ECOG 4 | 0 | 0
  Months 49-54: ECOG 5 | 0 | 0
  Months 55-60: number analyzed (Participants) | 19 | 0
  Months 55-60: Missing | 2 | 0
  Months 55-60: ECOG 0 | 11 | 0
  Months 55-60: ECOG 1 | 6 | 0
  Months 55-60: ECOG 2 | 0 | 0
  Months 55-60: ECOG 3 | 0 | 0
  Months 55-60: ECOG 4 | 0 | 0
  Months 55-60: ECOG 5 | 0 | 0
  Months 61-66: number analyzed (Participants) | 15 | 0
  Months 61-66: Missing | 1 | 0
  Months 61-66: ECOG 0 | 8 | 0
  Months 61-66: ECOG 1 | 6 | 0
  Months 61-66: ECOG 2 | 0 | 0
  Months 61-66: ECOG 3 | 0 | 0
  Months 61-66: ECOG 4 | 0 | 0
  Months 61-66: ECOG 5 | 0 | 0
  Months 67-72: number analyzed (Participants) | 14 | 0
  Months 67-72: Missing | 0 | 0
  Months 67-72: ECOG 0 | 8 | 0
  Months 67-72: ECOG 1 | 6 | 0
  Months 67-72: ECOG 2 | 0 | 0
  Months 67-72: ECOG 3 | 0 | 0
  Months 67-72: ECOG 4 | 0 | 0
  Months 67-72: ECOG 5 | 0 | 0
  Months 73-78: number analyzed (Participants) | 13 | 0
  Months 73-78: Missing | 0 | 0
  Months 73-78: ECOG 0 | 7 | 0
  Months 73-78: ECOG 1 | 5 | 0
  Months 73-78: ECOG 2 | 1 | 0
  Months 73-78: ECOG 3 | 0 | 0
  Months 73-78: ECOG 4 | 0 | 0
  Months 73-78: ECOG 5 | 0 | 0
  Months 79-84: number analyzed (Participants) | 10 | 0
  Months 79-84: Missing | 0 | 0
  Months 79-84: ECOG 0 | 6 | 0
  Months 79-84: ECOG 1 | 4 | 0
  Months 79-84: ECOG 2 | 0 | 0
  Months 79-84: ECOG 3 | 0 | 0
  Months 79-84: ECOG 4 | 0 | 0
  Months 79-84: ECOG 5 | 0 | 0
  Months 85-90: number analyzed (Participants) | 10 | 0
  Months 85-90: Missing | 0 | 0
  Months 85-90: ECOG 0 | 4 | 0
  Months 85-90: ECOG 1 | 5 | 0
  Months 85-90: ECOG 2 | 1 | 0
  Months 85-90: ECOG 3 | 0 | 0
  Months 85-90: ECOG 4 | 0 | 0
  Months 85-90: ECOG 5 | 0 | 0
  Months 91-96: number analyzed (Participants) | 9 | 0
  Months 91-96: Missing | 0 | 0
  Months 91-96: ECOG 0 | 5 | 0
  Months 91-96: ECOG 1 | 4 | 0
  Months 91-96: ECOG 2 | 0 | 0
  Months 91-96: ECOG 3 | 0 | 0
  Months 91-96: ECOG 4 | 0 | 0
  Months 91-96: ECOG 5 | 0 | 0
  Months 97-102: number analyzed (Participants) | 8 | 0
  Months 97-102: Missing | 2 | 0
  Months 97-102: ECOG 0 | 4 | 0
  Months 97-102: ECOG 1 | 2 | 0
  Months 97-102: ECOG 2 | 0 | 0
  Months 97-102: ECOG 3 | 0 | 0
  Months 97-102: ECOG 4 | 0 | 0
  Months 97-102: ECOG 5 | 0 | 0
  Months 103-108: number analyzed (Participants) | 5 | 0
  Months 103-108: Missing | 1 | 0
  Months 103-108: ECOG 0 | 1 | 0
  Months 103-108: ECOG 1 | 3 | 0
  Months 103-108: ECOG 2 | 0 | 0
  Months 103-108: ECOG 3 | 0 | 0
  Months 103-108: ECOG 4 | 0 | 0
  Months 103-108: ECOG 5 | 0 | 0
  Months 109-114: number analyzed (Participants) | 3 | 0
  Months 109-114: Missing | 0 | 0
  Months 109-114: ECOG 0 | 1 | 0
  Months 109-114: ECOG 1 | 2 | 0
  Months 109-114: ECOG 2 | 0 | 0
  Months 109-114: ECOG 3 | 0 | 0
  Months 109-114: ECOG 4 | 0 | 0
  Months 109-114: ECOG 5 | 0 | 0
  Months 115-120: number analyzed (Participants) | 3 | 0
  Months 115-120: Missing | 0 | 0
  Months 115-120: ECOG 0 | 2 | 0
  Months 115-120: ECOG 1 | 0 | 0
  Months 115-120: ECOG 2 | 1 | 0
  Months 115-120: ECOG 3 | 0 | 0
  Months 115-120: ECOG 4 | 0 | 0
  Months 115-120: ECOG 5 | 0 | 0
  Months 121-126: number analyzed (Participants) | 3 | 0
  Months 121-126: Missing | 0 | 0
  Months 121-126: ECOG 0 | 1 | 0
  Months 121-126: ECOG 1 | 1 | 0
  Months 121-126: ECOG 2 | 1 | 0
  Months 121-126: ECOG 3 | 0 | 0
  Months 121-126: ECOG 4 | 0 | 0
  Months 121-126: ECOG 5 | 0 | 0
  Months 127-132: number analyzed (Participants) | 3 | 0
  Months 127-132: Missing | 0 | 0
  Months 127-132: ECOG 0 | 1 | 0
  Months 127-132: ECOG 1 | 2 | 0
  Months 127-132: ECOG 2 | 0 | 0
  Months 127-132: ECOG 3 | 0 | 0
  Months 127-132: ECOG 4 | 0 | 0
  Months 127-132: ECOG 5 | 0 | 0
  Months 133-138: number analyzed (Participants) | 3 | 0
  Months 133-138: Missing | 0 | 0
  Months 133-138: ECOG 0 | 1 | 0
  Months 133-138: ECOG 1 | 2 | 0
  Months 133-138: ECOG 2 | 0 | 0
  Months 133-138: ECOG 3 | 0 | 0
  Months 133-138: ECOG 4 | 0 | 0
  Months 133-138: ECOG 5 | 0 | 0
  Months 139-144: number analyzed (Participants) | 3 | 0
  Months 139-144: Missing | 0 | 0
  Months 139-144: ECOG 0 | 1 | 0
  Months 139-144: ECOG 1 | 1 | 0
  Months 139-144: ECOG 2 | 1 | 0
  Months 139-144: ECOG 3 | 0 | 0
  Months 139-144: ECOG 4 | 0 | 0
  Months 139-144: ECOG 5 | 0 | 0
  Months 145-150: number analyzed (Participants) | 3 | 0
  Months 145-150: Missing | 0 | 0
  Months 145-150: ECOG 0 | 1 | 0
  Months 145-150: ECOG 1 | 1 | 0
  Months 145-150: ECOG 2 | 1 | 0
  Months 145-150: ECOG 3 | 0 | 0
  Months 145-150: ECOG 4 | 0 | 0
  Months 145-150: ECOG 5 | 0 | 0
  Months 151-156: number analyzed (Participants) | 3 | 0
  Months 151-156: Missing | 0 | 0
  Months 151-156: ECOG 0 | 1 | 0
  Months 151-156: ECOG 1 | 1 | 0
  Months 151-156: ECOG 2 | 1 | 0
  Months 151-156: ECOG 3 | 0 | 0
  Months 151-156: ECOG 4 | 0 | 0
  Months 151-156: ECOG 5 | 0 | 0
  Last available value: Missing | 9 | 0
  Last available value: ECOG 0 | 20 | 1
  Last available value: ECOG 1 | 25 | 0
  Last available value: ECOG 2 | 4 | 0
  Last available value: ECOG 3 | 1 | 0
  Last available value: ECOG 4 | 0 | 0
  Last available value: ECOG 5 | 5 | 0

ADVERSE EVENTS:
Time Frame: From signing the ICF in STEP until 30 days after the last sorafenib dose, with a mean duration of 26 months. Reporting for the numbers of all-cause mortality considers all deaths that occurred at any time during the study until the end of the follow up (with a mean duration of 26 months).
Groups:
- Sorafenib Monotherapy: Sorafenib monotherapy
- Sorafenib+Erlotinib: Sorafenib+Erlotinib
Arm/Group | Sorafenib Monotherapy | Sorafenib+Erlotinib
All-Cause Mortality (participants affected / at risk) | 62/203 | 0/1
Serious Adverse Events (participants affected / at risk) | 114/203 | 1/1
Other Adverse Events (participants affected / at risk) | 151/203 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Monotherapy (N=203) | Sorafenib+Erlotinib (N=1)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 3 (3) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (3) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neurological procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiocardiogram (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Monotherapy (N=203) | Sorafenib+Erlotinib (N=1)
Anaemia (Blood and lymphatic system disorders) | 15 (16) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (18) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (13) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 100 (147) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 12 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (10) | 0 (0)
Asthenia (General disorders) | 6 (7) | 0 (0)
Fatigue (General disorders) | 33 (41) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (9) | 0 (0)
Amylase increased (Investigations) | 9 (13) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 0 (0)
Haemoglobin decreased (Investigations) | 7 (9) | 0 (0)
Lipase increased (Investigations) | 13 (15) | 0 (0)
Platelet count decreased (Investigations) | 6 (6) | 0 (0)
Weight decreased (Investigations) | 10 (10) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (8) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (12) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 82 (96) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 16 (19) | 0 (0)
Flushing (Vascular disorders) | 3 (7) | 0 (0)
Hypertension (Vascular disorders) | 26 (26) | 1 (2)

LIMITATIONS AND CAVEATS:
No primary endpoints were defined specifically for study STEP as the primary purpose of this study was to enable patients to continue sorafenib treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not present or publish data until the full multi-center Trial has been reported in full. If a publication is not published within 24 [OR: 12-THIS IS MINIMUM] months after completion of the Trial, the PI may present or publish data.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT00625378/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT00625378/SAP_001.pdf